CLINICAL TRIAL: NCT05322174
Title: The Baby Care Study: Online Support for New Parents
Brief Title: The Baby Care Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Associate Professor of Pediatrics, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005999
Record Dates: First submitted 2022-03-28; First posted 2022-04-11 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Sleep; Parenting; Eating Behavior; Obesity
MeSH Terms: conditions — Feeding Behavior; Obesity | interventions — Infant Care

STUDY DESIGN:
Masking Description: Participants are randomly assigned to one of two online, behavioral interventions. Because the participants will know which behaviors are promoted to their group, and study staff will be interacting with the participants in their groups, masking is not possible. However, which group is considered the main intervention versus the attention control will not be known to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby Sleep (Experimental): Those randomized to this intervention group will receive an interactive online intervention focused on promoting infant sleep. This will include membership in a private Facebook group with support provided in the group, including weekly resources in the form of videos and tip sheets. To supplement this, they will also receive items meant to help with sleep (ex. sleep sack, baby sleep book).
  Interventions: Behavioral: Baby Sleep
- Baby Care (Active Comparator): The active control condition will parallel the intervention, but will be focused on general baby care and not sleep. Participants will be added to a private Facebook group in which general baby care information will be shared (e.g., bathing, play) and will receive items to help with general baby care (e.g., baby care kit with items such as nail clippers and comb; general baby care book). Topics related to sleep and feeding will not be highlighted in this group.
  Interventions: Behavioral: Baby Care

INTERVENTIONS:
Behavioral: Baby Sleep — See arm description
  Arms: Baby Sleep
Behavioral: Baby Care — See arm description
  Arms: Baby Care

SUMMARY:
The objective of this study is to provide pilot data on the feasibility and effectiveness of a web-based social networking intervention designed to promote sleep early in infancy and to explore the potential for this approach to promote healthy feeding routines, eating behaviors, and weight outcomes in subsequent larger-scale intervention research. First-time parents will be recruited (n=66) and randomized to an 8-week web-based social networking sleep intervention or general baby care control group with interventions beginning at infant age 8 weeks. Parents will complete online surveys, with research questions including: 1) whether the sleep intervention leads to longer nighttime and total sleep duration and decreased night waking among infants and 2) longer infant sleep bouts and improved parent sleep duration, stress, parenting efficacy, and parenting satisfaction. We will also examine infants' routines, feeding and eating behaviors, and emotion regulation to inform the application of this approach for childhood obesity prevention. The pilot research will provide insights into intervention feasibility, effects on infant sleep, and potential impacts on feeding and eating outcomes, informing our next steps.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking, first-time parents/legal guardians >18 years of a young infant who is < 6 weeks at the time of recruitment (or pregnant first-time parents expecting an infant soon). We will not include any parents who report that they do not have access to or an interest in using a private group on social media and/or online surveys.

Exclusion Criteria:

* We will exclude families not meeting age criteria, as well as any parents who report that they do not have access to or an interest in using a private group on social media and/or online surveys. We will also exclude parents of infants who are born premature (prior to 37 weeks gestational age) and parents of multiples (twins, triplets, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Nighttime infant sleep duration | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Total hours of nighttime sleep for the infant, from the Brief Infant Sleep Questionnaire (Sadeh)
Total infant sleep duration | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Total hours of sleep for the infant, from the Brief Infant Sleep Questionnaire (Sadeh)
Number of infant night wakings | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Number of night wakings for the infant, from the Brief Infant Sleep Questionnaire (Sadeh)

SECONDARY OUTCOMES:
Infant's longest sleep bout | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Longest sleep bout for the infant, item written by the study team
Parent sleep duration | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Total hours of sleep per night reported by the parent, from the Pittsburgh Sleep Quality Index (Buysse)
Parent stress | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Stress scores from the Perceived Stress Scale (Cohen) (minimum value = 0, maximum value = 40; higher scores mean more stress)
Parenting self-efficacy | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Efficacy scale from the Parenting Sense of Competence Questionnaire (Gibaud-Wallston & Wandersman)
Parenting satisfaction | From baseline (infant age 6 weeks) to follow-up (age 7 months)
  Satisfaction scale from the Parenting Sense of Competence Questionnaire (Gibaud-Wallston & Wandersman)

OTHER OUTCOMES:
Infant routines | Mid-point (infant age 3 months) to post-test (infant age 4 months)
  Routine subscale from the Infant Parenting Styles Questionnaire (Arnott & Brown)
Limit exposure | Follow-up (infant age 7 months)
  Limit exposure subscale from the Structure & Control in Parent Feeding Questionnaire (Savage)
Mealtime routines | Follow-up (infant age 7 months)
  Mealtime routines subscale from the Structure & Control in Parent Feeding Questionnaire (Savage)
Restriction | Follow-up (infant age 7 months)
  Restriction subscale from the Structure & Control in Parent Feeding Questionnaire (Savage)
Pressure to eat | Follow-up (infant age 7 months)
  Pressure to eat subscale from the Structure & Control in Parent Feeding Questionnaire (Savage)
Nutritional quality | Follow-up (infant age 7 months)
  We will create a composite variable that is a proxy for nutritional quality using the frequencies that the consumption of various food groups (vegetables, fruit, fried food, sweets) are reported
Emotion regulation | Follow-up (infant age 7 months)
  Regulation superfactor from the Infant Behavior Questionnaire Very Short Form (Rothbart)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Anzman-Frasca S, Goldsmith J, Hassinger AB, Wilding G, Buxton OM, Savage JS. Exploring Effects of a Randomized Online Infant Sleep Intervention on Weight-Related Outcomes Into Toddlerhood. Obesity (Silver Spring). 2025 Oct 26. doi: 10.1002/oby.70037. Online ahead of print. PMID 41140015
- [Derived] Anzman-Frasca S, Goldsmith J, Hassinger AB, Savage JS, Gupta V. Implementation and Effects of an Online Intervention Designed to Promote Sleep During Early Infancy: A Randomized Trial. Nat Sci Sleep. 2025 May 24;17:1037-1048. doi: 10.2147/NSS.S501807. eCollection 2025. PMID 40438635